CLINICAL TRIAL: NCT07242508
Title: Efficacy of a New Infant Formula Composition on Gut Health in Infants: A Prospective Randomized Double-blind Placebo-controlled Trial
Brief Title: Efficacy of a New Infant Formula Composition on Gut Health in Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ECCT2831
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Infants
Keywords: infant; formula; microbiota; gut health; RCT
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental infant formula (Experimental): Infant formula with bioactive ingredients
  Interventions: Other: Infant Formula with bioactive ingredients
- Control formula (Placebo Comparator): Standard infant formula
  Interventions: Other: Infant Formula

INTERVENTIONS:
Other: Infant Formula — ad-libitum consumption of infant formula
  Arms: Control formula
Other: Infant Formula with bioactive ingredients — ad-libitum consumption
  Arms: Experimental infant formula

SUMMARY:
The aim of this study is to investigate potential health benefits of the experimental formula. The main objective is whether the experimental formula elevates the relative abundance of Bifidobacterium in stool samples after 10 weeks, as compared a standard formula, aka control formula. In addition other markers of gut health, such as stool characteristics, and gut health symptoms will be monitored

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full term, infants with a birth weight between 2500-4500 grams
* Parents independently from study decided to not breastfeed their infant
* Parents agree to feed the assigned study formula as the infant's sole source of nutrition for the duration of the study
* have read and voluntarily signed an informed consent form
* parents are capable of completing study procedures required by the protocol

Exclusion Criteria:

* suffering from any anatomic and/or physiologic condition that would interfere with normal growth, development or feeding
* are required to take medications or supplements known to influence growth and development
* have a maternal history with known adverse effects on the fetus and/or the newborn infant
* have previous or current antibiotics use (antibiotics administered during delivery are permitted)
* have received or are planning to receive probiotics, prebiotics, or nutritional supplements prior to and throughout the trial (excluding vitamin D and vitamin K supplementation)
* personal history of or parents/siblings diagnosed with cow's milk protein allergy or lactose intolerance
* multiple birth
* participation in another trial

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Bifidobacterium | From enrollment to the end of treatment at 10 weeks
  Relative abundance of bifidobacterium from stool samples

IPD SHARING:
Plan to Share IPD: No